CLINICAL TRIAL: NCT00332241
Title: A Multicenter Double-Blind, Randomized, Placebo-Controlled, Flexible-Dosed, Parallel-Group Study of Aripiprazole Flexibly Dosed in the Treatment of Children and Adolescents With Autistic Disorder (AD)
Brief Title: Study of Aripiprazole in the Treatment of Children and Adolescents With Autistic Disorder (AD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-178
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Results first posted 2009-07-23 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Autistic Disorder
Keywords: Serious behavioral problems in children and adolescents with AD; Behavioral Problems
MeSH Terms: conditions — Autistic Disorder; Problem Behavior | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Experimental): Active Abilify
  Interventions: Drug: Aripiprazole
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 5, 10, or 15 mg, once daily, 8 weeks
  Other Names: Abilify
  Arms: A1
Drug: Placebo — Tablets, Oral, once daily, 8 weeks
  Arms: A2

SUMMARY:
This study will compare the effectiveness (how well the drug works) of aripiprazole, flexibly dosed with a placebo, in reducing serious behavioral problems in children and adolescents with a diagnosis of autistic disorder (AD).

ELIGIBILITY:
Inclusion Criteria:

* Meets current Diagnostic and Statistical Manual for Mental Disorders-Fourth Edition (DSM-IV) diagnostic criteria for AD and demonstrates serious behavioral problems. Diagnosis confirmed by Autism Diagnostic Interview- Revised (ADI-R)
* CGI score > = 4 AND and Aberrant Behavior Checklist (ABC) Irritability/Agitation subscale score > = 18 at screening and baseline (randomization)
* Mental age of at least 18 months
* Male or female 6 to 17 years of age, inclusive, at the time of randomization

Exclusion Criteria:

* Patients considered treatment resistant to neuroleptic medication based on lack of therapeutic response to 2 different neuroleptics after treatment of at least 3 weeks each.
* Patients previously treated and not responding to aripiprazole treatment
* The patient is currently diagnosed with another disorder on the autism spectrum, including PDD-NOS, Asperger's Disorder, Rett's Disorder, Fragile-X Syndrome or Childhood Disintegrative Disorder
* Current diagnosis of bipolar disorder, psychosis, or schizophrenia, or major depression
* A seizure in the past year
* History of severe head trauma or stroke
* Patients undergoing non-pharmacologic therapies (e.g., psychotherapy, behavioral modification) must have started at least 2 months prior to the initial screening visit and must remain in a consistent treatment program for the duration of the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (9):
  - Marsella, Gregory, Boca Raton, Florida
  - Child Neurology Associates, Pc, Atlanta, Georgia
  - University Of Louisville, Louisville, Kentucky
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Center For Psychiatry And Behavioral Medicine, Las Vegas, Nevada
  - Suny - Stony Brook School Of Medicine, Stony Brook, New York
  - Univ Of Nc, Chapel Hill, North Carolina
  - Ut Medical Group, Memphis, Tennessee
  - Red Oak Psychiatry Associates, Pa, Houston, Texas

REFERENCES:
- [Background] Owen R, Sikich L, Marcus RN, Corey-Lisle P, Manos G, McQuade RD, Carson WH, Findling RL. Aripiprazole in the treatment of irritability in children and adolescents with autistic disorder. Pediatrics. 2009 Dec;124(6):1533-40. doi: 10.1542/peds.2008-3782. PMID 19948625
- [Derived] Mankoski R, Stockton G, Manos G, Marler S, McQuade R, Forbes RA, Marcus R. Aripiprazole treatment of irritability associated with autistic disorder and the relationship between prior antipsychotic exposure, adverse events, and weight change. J Child Adolesc Psychopharmacol. 2013 Oct;23(8):572-6. doi: 10.1089/cap.2012.0075. PMID 24138011
- [Derived] Robb AS, Andersson C, Bellocchio EE, Manos G, Rojas-Fernandez C, Mathew S, Marcus R, Owen R, Mankoski R. Safety and tolerability of aripiprazole in the treatment of irritability associated with autistic disorder in pediatric subjects (6-17 years old):results from a pooled analysis of 2 studies. Prim Care Companion CNS Disord. 2011;13(1):PCC.10m01008. doi: 10.4088/PCC.10m01008gry. PMID 21731831
- [Derived] Aman MG, Kasper W, Manos G, Mathew S, Marcus R, Owen R, Mankoski R. Line-item analysis of the Aberrant Behavior Checklist: results from two studies of aripiprazole in the treatment of irritability associated with autistic disorder. J Child Adolesc Psychopharmacol. 2010 Oct;20(5):415-22. doi: 10.1089/cap.2009.0120. PMID 20973712

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: oral placebo once daily (QD)
- Aripiprazole: oral aripiprazole 2 to 15 mg QD
Period: Overall Study
Arm/Group | Placebo | Aripiprazole
Started | 51 | 47
Completed | 36 | 39
Not Completed | 15 | 8
Not completed — Lack of Efficacy | 6 | 1
Not completed — Adverse Event | 3 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aripiprazole | Total
Number analyzed (Participants) | 51 | 47 | 98
Age, Customized [Number; unit: participants]
  6 to 12 years | 46 | 37 | 83
  13 to 17 years | 5 | 10 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 44 | 42 | 86
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 11 | 18
  White | 41 | 32 | 73
  Other | 3 | 1 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 8 | 6 | 14
  Not Hispanic/Latino | 43 | 41 | 84
Weight Group [Number; unit: Participants]
  <40 kilograms | 32 | 26 | 58
  ≥40 kilograms | 19 | 21 | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/cm2] | 19.96 (5.392) | 21.08 (5.394) | 20.50 (5.395)
Height [Mean (Standard Deviation); unit: centimeters] | 138.6 (14.7) | 140.9 (18.80) | 139.7 (16.74)
Weight [Mean (Standard Deviation); unit: kilograms] | 40.6 (18.92) | 43.9 (19.15) | 42.2 (19.01)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (Week 8 - Baseline) in the Autistic Behavior Checklist (ABC) Irritability Subscale Score
Description: The ABC is a 58-item informant-based assessment of problem behaviors in children/adolescents with mental retardation. Items are rated on a 4-point scale (0=no problem, 3=severe problem), and resolve into 5 domain subscales. A decrease in score indicates improvement.
Time Frame: Week 8
Population: Efficacy population=all randomized participants minus 2 patients in the placebo group (1 lost to follow-up, 1 withdrew consent) and 1 participant in the aripiprazole group who discontinued due to AE on Day 2. Data set is LOCF.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 49 | 46
units on a scale | -5.0 (1.43) | -12.9 (1.44)

2. Secondary Outcome: Mean Clinical Global Impressions Improvement Scale (CGI-I) Score
Description: The CGI scale is a clinician-rated global assessment of a patient's improvement over time. Baseline assessment rated a patient's condition on a 7-point scale (1=no symptoms, 7=very severe symptoms). Subsequent assessed improvement relative to baseline symptoms on a 7-point CGI-I item scale (1=very much improved, 7=very much worse).
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 49 | 46
units on a scale | 3.6 (0.18) | 2.2 (0.18)

3. Secondary Outcome: Number of Participants With Response at Week 8
Description: Response defined as a ≥ 25% reduction from baseline to endpoint in the ABC Irritability Subscale score and a CGI-I score of 1 or 2 at endpoint
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 49 | 46
participant | 7 | 24

4. Secondary Outcome: Mean Change (Week 8 - Baseline) in the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS; Compulsion Scale Only)
Description: CY-BOCS=10-item assessment of obsessive-compulsive symptoms in patients <18 years. 5 items pertaining to compulsions rate symptoms (time spent, interference with functioning, distress, resistance, control) on a 5-point scale (0=no symptoms/minimum severity, 4=extreme symptoms/maximum severity). A decrease in value indicates improvement.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 44 | 43
units on a scale | -0.8 (0.52) | -3.8 (0.50)

5. Secondary Outcome: Mean Change (Week 8 - Baseline) in the Other ABC Subscale Scores
Description: Mean change (Week 8 - baseline) in the other ABC subscale scores (lethargy/social withdrawal; stereotypic behavior; hyperactivity/ noncompliance; inappropriate speech). A decrease in value indicates improvement
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units of a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 49 | 46
units of a scale
  ABC Hyperactivity Subscale Score | -2.8 (1.5) | -12.7 (1.52)
  ABC Stereotypy Subscale Score | -2.0 (0.62) | -4.8 (0.63)
  ABC Inappropriate Speech Subscale Score | -0.4 (0.39) | -2.5 (0.39)
  ABC Social Withdrawal Subscale Score | -6.2 (1.13) | -7.9 (1.15)

6. Secondary Outcome: Mean Change (Week 8 - Baseline) in CGI-Severity (CGI-S)
Description: A CGI-S assessment (a 7-point scale to evaluate the severity of symptoms) was performed at baseline (1=no symptoms; 7=very severe symptoms). The patient's improvement relative to the symptoms at baseline on were assessed on a 7-point CGI-I (1=very much improved; 7=very much worse). A decrease in value indicates improvement.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 40 | 40
units on a scale | -0.4 (0.15) | -1.2 (0.14)

7. Secondary Outcome: Summary of Safety
Description: Deaths, Adverse Events (AEs), Serious AEs (SAEs), Treatment-Emergent AEs and AEs leading to discontinuation
Time Frame: continuous throughout the study
Population: Safety population=all randomized participants minus 1 patient in the placebo group lost to follow-up. Data set is LOCF.
Measure: Number; unit: participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 50 | 47
participants
  Deaths | 0 | 0
  Treatment-emergent SAEs | 0 | 0
  AEs leading to discontinuation | 3 | 5
  Treatment-emergent AEs overall | 36 | 43
  Treatment-emergent AEs realted to study drug | 25 | 39
  Treatment-emergent extrapyramidal symptom AEs | 4 | 7

8. Secondary Outcome: Change From Baseline in Body Weight
Description: Adjusted mean change (Week 8 - baseline) in body weight
Time Frame: Week 8
Population: Safety population=all randomized participants minus 1 patient in the placebo group lost to follow-up. Includes all participants with weight measurement at baseline and timepoint. Data set is LOCF.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 49 | 45
kilograms | 0.8 (0.29) | 2.0 (0.30)

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 38/47 | 29/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=47) | Placebo (N=50)
INSOMNIA (Psychiatric disorders) | 3 | 4
AGGRESSION (Psychiatric disorders) | 1 | 4
TREMOR (Nervous system disorders) | 4 | 0
DROOLING (Nervous system disorders) | 4 | 0
HEADACHE (Nervous system disorders) | 3 | 8
SEDATION (Nervous system disorders) | 5 | 1
SOMNOLENCE (Nervous system disorders) | 8 | 2
VOMITING (Gastrointestinal disorders) | 7 | 2
DIARRHOEA (Gastrointestinal disorders) | 4 | 5
NASOPHARYNGITIS (Infections and infestations) | 2 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 5
ENURESIS (Renal and urinary disorders) | 3 | 4
INCREASED APPETITE (Metabolism and nutrition disorders) | 7 | 5
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 1
FATIGUE (General disorders) | 10 | 2
PYREXIA (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.